CLINICAL TRIAL: NCT06240832
Title: Aerobic Capacity Muscle Strength and Health Related Quality of Life in Children With Chronic Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ibrahim, assistant lecturer, pediatric department of physical therapy,principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P. T. REC/012/003479
Record Dates: First submitted 2024-01-07; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Chronic Liver Failure
Keywords: aerobic capacity; chronic liver disease; muscle strength
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Intervention Model Description: One group of children ages more than 6ys will recruited and assessed pre and post of study completion for 12week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic and strength training in children with CLD (Experimental): AEROBIC AND STRENGTHENING EXERCISE USING TREADMILL AND WEIGHT TO IMPROVE FUNCTIONAL OUTCOMES IN CHILDREN WITH CHRONIC LIVER DISEASE
  Interventions: Other: Physical therapy exercise

INTERVENTIONS:
Other: Physical therapy exercise — Endurance, strength and stretching training in Chronic liver disease children
  Other Names: Designated physical therapy program

SUMMARY:
Physical therapy program for children with chronic liver disease consist of gait training, strengthening ex for UL&ll, stretching exercise to improve physical fitness and quality of life

DETAILED DESCRIPTION:
Intervention study for one group of children diagnosed with chronic liver disease ages more than 6ys, study include assessment and intervention, assessment of 6MWt, grip strength by hand held dynamometer, quadriceps strength by Lafayette, al children subjected to laboratory investigation pre and post of study completion, anthropometric measure, quality of life and fatigue assessment then all children will perform physical therapy program of gait training muscle strengthening for 8 week

ELIGIBILITY:
Inclusion Criteria:

* Their age ranged from7 to14 years old.
* Residence in Cairo to be able to attend the rehabilitation program.
* Diagnosis of CLD as (Wilson disease, autoimmune hepatitis, chronic cholestasis , ….etc).
* All children were medically stabled
* All children had the same socioeconomic status

Exclusion Criteria:

* Complication that prevent children from performing maximal exercise test as fracture of both upper and lower limbs, cardiovascular instability and muscle disease in patient with glycogen storage disease(GSD) or abnormal creatine phosphokinase(CPK).
* Patients with cognitive and motor disorders as in case of hepatic encephalopathy and or ascites.
* Patients who underwent liver transplantation.
* Patient with end stage liver disease.
* History of variceal bleeding from one month ago or less.
* No other system disease (chest, cardiac and nervous system).
* Medical examination no hernia.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
aerobic capacity | 8week
  it was assessed by 6 minute walk test(6-MWT) in meter, The distance in meters was recorded at the end of the six minutes.
grip strength | 8week
  it was assessed by pneumatic hand held dynamometer ,was measured in pounds per square inch (PSI). The child was sitting on a chair with or without arm rest, back supported, and both feet rested on the floor. The right arm was beside the body, with adducted shoulder, elbow flexed 90°, forearm in neutral position, wrist from 0° to 30° extension, and 0° to 15° of ulnar deviation. Child was instructed to hold and compress the pneumatic handle of dynamometer as much strength as possible with the tested hand
quadriceps strength | 8 week
  it was assessed by Lafayette hand held dynamometer(LHHD)Child position was sitting on chair with back straight, hip and knee were in 90-degree flexion. LHHD was fixed on distal third of anterior surface of child leg while his/her tested thigh was stabilizing and then the child was instructed to perform maximal isometric knee extension and hold for 6 sec against LHHD sensor pad.
health related quality of life | 8week
  The Arabic version of child self-report Pediatric Quality of Life Inventory core scale version 4 (PedsQI) was used to assess HRQOL. PedsQI core scale designed to measure HRQOL in children and adolescents ages from 2 to18years. Each item of the questionnaire rated based on a rating scale from 0-4. Then, each item score was linearly converted on assessment scale from 0 to 100;0=100, 1=75, 2=50, 3=25, 4=0 then overall score calculated for all domains through dividing all answered items over whole number of items, with higher scores indicate a better HRQOL
fatigue | 8 weeks
  It was assessed by the PedsQI multidimensional fatigue scale version 3. It is composed of 3 domains; general fatigue, sleep/rest fatigue and cognitive fatigue,Each item score converted on a scale from 0 to 100: 0=100, 1=75, 2=50, 3=25, 4=0 then overall score calculated for all domains through dividing all answered items over whole number of items, with higher scores indicate lower level of fatigue

SECONDARY OUTCOMES:
hemoglobin | 8week
  A blood sample was taken for complete blood count (CBC )hemoglobin
liver enzymes | 8week
  A blood sample was taken for liver enzymes (Total bilirubin ,Direct bilirubin ) unit of measure (mg/dl)
minerals | 8week
  A blood sample was taken for minerals concentration (sodium Na,potassium K, magnissium M, calciumCa, posphorus P and create) unit of measure (mmol/l)
mid upper arm circumference in centimeter | 8 weeks
  assessed by tape measure,the tape was passed around the arm at the mid-point of the upper right arm halfway between the acromion process and the olecranon process
triceps skin fold thickness | 8 weeks
  it was assessed by holtain skinfold calipers in millimeter
height in meter (m) | 8 weeks
  assessed by stadiometre
weight in kilogrms (Kg) | 8 weeks
  assess by electronic scale
body mass index | 8weeks
  height/weight kg/m2
mid upper muscle circumference | 8weeks
  assessed by calculators that substract triceps skin fold thickness from mid upper arm circumference
mid upper leg circumference in centimetre | 8 weeks
  assessed by tape measure at mid -point between iliac crest and mid of patella

CONTACTS AND LOCATIONS:
Overall Officials: Heba A IBRAHIM, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

REFERENCES:
- [Result] Zenith L, Meena N, Ramadi A, Yavari M, Harvey A, Carbonneau M, Ma M, Abraldes JG, Paterson I, Haykowsky MJ, Tandon P. Eight weeks of exercise training increases aerobic capacity and muscle mass and reduces fatigue in patients with cirrhosis. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1920-6.e2. doi: 10.1016/j.cgh.2014.04.016. Epub 2014 Apr 24. PMID 24768811